CLINICAL TRIAL: NCT02579473
Title: A Multi-center, Open-label, Multiple Ascending Dosage-ranging Cohort (MAD) Study in Early, Untreated or Stably Treated Subjects With Parkinson's Disease (PD), to Determine the Safety, Tolerability and Pharmacokinetics (PK) of Injections of SER-214 Administered Subcutaneously Once a Week for Two Weeks After 0-2 Weeks of Dose Titration
Brief Title: A Study of Weekly Subcutaneous Injections of SER-214 in Subjects With Parkinson's Disease (PD), to Determine the Safety, Tolerability and Pharmacokinetic (PK) Profile of SER-214
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Serina Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SER-214 Ia
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2022-10

CONDITIONS: Parkinson's Disease
Keywords: Continuous dopaminergic stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 0 (Experimental): Subjects in Cohort 0 will receive a single subcutaneous injection of 20 mg SER-214, followed by a two week wash-out period, to determine safety, tolerability and PK and terminal "wash-out" of rotigotine and pro-drug SER-214.
  Interventions: Drug: SER-214
- Cohort 1 (Experimental): Subjects in Cohort 1 will receive a single SC injection of 50 mg SER-214 at the beginning of each week for two consecutive weeks, followed by a two week wash-out period, to determine safety, tolerability and PK and terminal "wash-out" of rotigotine and pro-drug SER-214.
  Interventions: Drug: SER-214
- Cohort 2 (Experimental): Subjects in Cohort 2 will receive a single SC injection of 50 mg SER-214 at the beginning of week one, followed by a weekly SC injection of 100 mg SER-214 for two consecutive weeks, followed by a two week wash-out period, to determine safety, tolerability and PK and terminal "wash-out" of rotigotine and pro-drug SER-214.
  Interventions: Drug: SER-214
- Cohort 3 (Experimental): Subjects in Cohort 3 will receive a single SC injection of 50 mg SER-214 at the beginning of week one, followed by a single SC injection of 100 mg SER-214 at the beginning of week two, followed by a single SC injection of 200 mg SER-214 for two consecutive weeks, followed by a two week wash-out period, to determine PK and terminal "wash-out" PK of rotigotine and pro-drug SER-214.
  Interventions: Drug: SER-214

INTERVENTIONS:
Drug: SER-214 — SER-214 is a poly(2-ethyl-oxazoline) (POZ) polymer conjugate of the potent dopamine agonist rotigotine that is designed to provide continuous drug delivery following a single weekly injection
  Other Names: POZ-rotigotine

SUMMARY:
SER-214 is a poly (2-ethyl-2oxazoline)(POZ) polymer conjugate of rotigotine, a potent dopamine agonist that has high affinity for the subclass of dopamine receptors in the brain that mediate dopamine signaling. SER-214 will be administered subcutaneously once a week via a standard 1 mL insulin syringe to determine the safety, tolerability and pharmacokinetic (PK) profile of released rotigotine and POZ-conjugate. Subjects in this study are eligible if they have early, stable or untreated Parkinson's disease and are still experiencing motor fluctuations.

DETAILED DESCRIPTION:
Clinical evidence suggests that dopamine agonists should be considered as an initial or early symptomatic therapy for PD. Current information indicates that the early use of long-acting dopaminergic agonists may protect against the development of motor complications by stimulating dopamine receptors in a non-pulsatile manner and by delaying the introduction of levodopa. In pre-clinical primate studies, L-dopa (short-acting, pulsatile) and dopaminergic agonists (long-acting; non pulsatile) provide comparable clinical benefit but with agonists inducing significantly less dyskinesia.

Chronic L-dopa treated animals develop gene changes that are associated with abnormal neuronal firing patterns and dyskinesias which are not seen with long-acting dopamine agonists. Based on pre-clinical and clinical study results, treatment of Parkinson's patients with long-acting levodopa or dopamine agonists should provide symptomatic benefit, and significantly delay the onset of motor complications. This can be accomplished with duodopa or continuous sc apomorphine but these treatments are associated with significant side effects. To date, no practical method of providing continuous drug delivery using a dopaminergic agent for therapy of patients with early PD to prevent the development of motor complications has been advanced through clinical trials.

SER-214 is being developed as a weekly sc injection that provides prompt onset of dopaminergic stimulation. Continuous levels of released rotigotine within the therapeutic window for relief of motor fluctuations have been observed in MPTP-treated cynomolgus macaques. PK determinations in normal monkeys for up to 13 weeks of treatment show that weekly injections of SER-214 provide continuous drug delivery of released plasma rotigotine within a predictable therapeutic range.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects 40-80 years of age inclusive
2. A diagnosis of idiopathic Parkinson's disease (PD) consistent with UK brain bank criteria
3. De novo PD patients and those on a stable regimen of anti-Parkinson's drugs for at least 4weeks prior to screening including anticholingerics, amantadine, MAO-B inhibitors, COMT inhibitors or levodopa, but not dopamine agonists
4. Free of clinically significant motor complications as determined by the investigator
5. Ability to complete up to four weeks of dosing once per week with two weeks of terminal "wash-out" PK
6. Ability to return to the clinic for blood sampling, clinical and laboratory assessment on scheduled days, based upon cohort
7. Mini Mental State Exam (MMSE) > 26
8. Women of child-bearing potential (WOCBP) must use a reliable method of contraception (e.g., oral contraceptive or long-term injectable or implantable hormonal contraceptive, double-barrier methods [such as condom plus diaphragm, condom plus spermicidal foam, condom plus sponge], or intra-uterine devices), and must have a negative serum pregnancy test at Screening and negative urine pregnancy test at baseline
9. Willing and able to comply with the study requirements including follow-up
10. Provide written informed consent
11. Cognitively intact sufficient to understand and provide informed consent
12. Approved by a central Eligibility Monitoring Committee (EMC) confirmed by EMC signature on the Enrollment Authorization Form (EAF)

Exclusion Criteria:

1. Subject has previously participated in this study.
2. Myocardial infarction within the past six months from screening
3. Ischemic stroke or transient ischemic event within the past two years from screening
4. Known sensitivity to dopamine agonists including nausea/vomiting, orthostatic hypotension, excessive sleep or impulse control disorder
5. Any major organ disease that substantially impairs life expectancy
6. History of cancer, other than basal cell carcinoma, within the past 10 years or subjects with any laboratory or physical exam or diagnostic procedure finding suggestive of current malignancy
7. Subjects who are known to be immunosuppressed or are receiving chronic treatment with immunosuppressive drugs
8. Subject with an atypical or secondary Parkinsonian (e.g., due to drugs, metabolic neurogenetic disorders, encephalitis, cerebrovascular disease or degenerative disease)
9. Any clinically significant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the Investigator, makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
10. Subject has moderate renal impairment (creatine > 2.5)
11. Subject has moderate (Child-Pugh categorization B, score 7-9) or severe (Child-Pugh categorization C, score 10-15) hepatic impairment.
12. Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (CSSRS) at Screening
13. Subject has known hypersensitivity to rotigotine or to any components or excipients of the study drug
14. Subject has a history of psychosis or hallucinations within the previous 12 months
15. Subject has received an investigational drug within 30 days of screening or is currently participating in an investigational drug or investigational device trial
16. Subject, who, for any reason, is judged by the Investigator to be inappropriate for this study, including a subject who is unable to communicate or cooperate with the Investigator or who has/had a clinically significant illness or abnormal physical examination that may compromise safety of the subject during the trial or affect ability of the subject to adhere to study procedures

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events and Serious Adverse Events | From initial sc dose of SER-214 up to six weeks of follow-up
  Change from Screening in frequency of adverse events (AEs) and serious adverse events (SAEs) at the Final Safety Visit
Percentage of patients in each cohort who discontinued therapy due to any adverse events {Tolerability} | From initial sc dose of SER-214 up to six weeks of follow-up
  Percentage of patients in each cohort who discontinued therapy due to any adverse events will be used as an assessment of tolerability
Safety - Vital Signs | From initial sc dose of SER-214 up to six weeks of follow-up
  Change from Screening in assessment of vital signs (pulse, blood pressure) at each study visit and Final Safety Visit
Safety - Abnormal Laboratory Results | From initial sc dose of SER-214 up to six weeks of follow-up
  Change from Screening in number of participants with laboratory test values of potential clinical importance
Safety - Treatment-Emergent Adverse Events | From initial sc dose of SER-214 up to six weeks of follow-up
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] will be assessed by the investigator (Yes/No).
Safety - ECG Changes | From initial sc dose of SER-214 up to six weeks of follow-up
  Change from Screening in assessment of electrocardiogram (ECG) parameters at each injection visit

SECONDARY OUTCOMES:
Fluctuation index | On injection days plasma samples will be taken at time 0, 1, 2, 4 and 8 hours
  On injection days plasma samples will be taken at time 0 (baseline), 1, 2, 4 and 8 hours post injection. PK samples will be used to determine (a) released plasma rotigotine and (b) total SER-214. PK data will be used to determine the Fluctuation Index
Maximum plasma concentration [C(max)] | On injection days plasma samples will be taken at time 0, 1, 2, 4 and 8 hours
  PK samples will be used to determine (a) released plasma rotigotine and (b) total SER-214. PK data will be used to determine the C(max)
Time to maximum concentration [T(max)] | On injection days plasma samples will be taken at time 0, 1, 2, 4 and 8 hours
  PK samples will be used to determine (a) released plasma rotigotine and (b) total SER-214. PK data will be used to determine the T(max)
Dose-adjusted area under the curve (AUC) | On injection days plasma samples will be taken at time 0, 1, 2, 4 and 8 hours
  PK samples will be used to determine (a) released plasma rotigotine and (b) total SER-214. PK data will be used to determine the dose-adjusted AUC
Unified Parkinson's Disease Rating Scale | From Screening up to six weeks of follow-up
  The UPDRS total (Parts I, II and III) will be determined at each study site visit and the Final Safety Visit
Unified Parkinson's Disease Rating Scale - Motor Part III Only | From Screening up to six weeks of follow-up
  The Motor UPDRS (Part III) will be determined as a separate outcome measure at each injection day visit
Epworth Sleepiness Scale (ESS) | From Screening up to six weeks of follow-up
  The ESS will be determined at Screening, first Follow-up visit, Final Safety Visit and any unscheduled visit to determine if escalating doses of SER-214 are associated with increase in somnolence
Columbia Suicide Severity Rating Scale (C-SSRS) | From Screening up to six weeks of follow-up
  The C-SSRS will be determined at Screening and Final Safety Visit and any unscheduled visit. C-SSRS assessed whether participant experienced following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Questionnaire for Impulsive-Compulsive Disorders in Parkinson's disease (QUIP) | From screening up to six weeks of follow-up
  The QUIP will be assessed at Screening and on the Final Safety Visit and any unscheduled visit to determine if there is any association between Impulsive-Compulsive behavior and SER-214 dose

CONTACTS AND LOCATIONS:
Overall Officials: David G Standaert, MD, PhD, Principal Investigator — Univeristy of Alabama-Birmingham School of Medicine, Division of Neurology
Locations (4):
- United States (4):
  - University of Alabama Birmingham, Birmingham, Alabama
  - MD Clinical, Hallandale, Florida
  - Georgia Regents University, Augusta, Georgia
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Eskow Jaunarajs KL, Standaert DG, Viegas TX, Bentley MD, Fang Z, Dizman B, Yoon K, Weimer R, Ravenscroft P, Johnston TH, Hill MP, Brotchie JM, Moreadith RW. Rotigotine polyoxazoline conjugate SER-214 provides robust and sustained antiparkinsonian benefit. Mov Disord. 2013 Oct;28(12):1675-82. doi: 10.1002/mds.25625. Epub 2013 Sep 3. PMID 24014074